CLINICAL TRIAL: NCT05489627
Title: Medial Collateral Ligament Reconstruction With Anteromedial Reinforcement for Medial and Anteromedial Rotatory Knee Instability
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Artromedical Konrad Malinowski Clinic (Other)
Responsible Party: Principal Investigator, Konrad Malinowski MD, Principal Investigator Konrad Malinowski MD, Artromedical Konrad Malinowski Clinic, Artromedical Konrad Malinowski Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-pro-ar-2022
Record Dates: First submitted 2022-08-03; First posted 2022-08-05 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Collateral Ligament, Knee; Sprain (Strain), Medial; Anterior Cruciate Ligament Injuries
MeSH Terms: conditions — Sprains and Strains; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: Single Group: Clinical trials with a single arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm of the study (Experimental): Medial knee instabilities will be addressed in this arm. Due to the fact that isolated injury of medial stabilizers of the knees is very rare, included will be patients with D concomitant ACL QTB reconstruction and MCL reconstruction. Any accompanying intraarticular injuries such as meniscal lesions will be addressed as well.
  17 patients will be included in this arm - this number was calculated and rounded up as a mean of number patients from studies of Alm et al. 2021 (17 patients in ACLR+MCLR group), Lee et al. 2020 (10 patients in ACLR+MCLR group), Kitamura et al. 2013 (16 patients in ACLR+MCLR group), LaPrade et al. 2012 (8 patients in ACLR+MCLR group), Lind et al. 2009 (34 patients in ACLR+MCLR group) and Kim et al. 2008 (12 patients in ACLR+MCLR group). All above referenced studies apart from the study of LaPrade et al. were retrospective.
  Interventions: Procedure: Medial Collateral Ligament Reconstruction With Anteromedial Reinforcement

INTERVENTIONS:
Procedure: Medial Collateral Ligament Reconstruction With Anteromedial Reinforcement — Medial knee instabilities will be addressed in this arm as described in the published technique: K. Malinowski, K. Hermanowicz, A. Góralczyk, R.F. LaPrade, Medial Collateral Ligament Reconstruction With Anteromedial Reinforcement for Medial and Anteromedial Rotatory Instability of the Knee, Arthrosc. Tech. 8 (2019) e807-e814. https://doi.org/10.1016/j.eats.2019.03.019.
  Due to the fact that isolated injury of medial stabilizers of the knees is very rare, included will be patients with concomitant ACL QTB reconstruction and abovedescribed MCL reconstruction. Any accompanying intraarticular injuries such as meniscal lesions will be addressed as well.

SUMMARY:
The aim of this study is to assess the outcomes of the combined quadriceps tendon-bone (QTB) ACLR and MCLR with anteromedial reinforcement performed as described in the published technique: K. Malinowski, K. Hermanowicz, A. Góralczyk, R.F. LaPrade, Medial Collateral Ligament Reconstruction With Anteromedial Reinforcement for Medial and Anteromedial Rotatory Instability of the Knee, Arthrosc. Tech. 8 (2019) e807-e814. https://doi.org/10.1016/j.eats.2019.03.019.

DETAILED DESCRIPTION:
Medial collateral ligament (MCL) injuries are one of the most common sports knee injuries, commonly occuring together with anterior cruciate ligament (ACL) injuries. Their effect on the knee joint can be detrimental with patients experiencing medial instability and anteromedial rotatory instability (AMRI), leading to progressive damage of the intraarticular structures. While healing potential of medial knee stabilizing structures is relatively high, medial collateral ligament reconstruction (MCLR) is sometimes indicated. Multiple reconstructions techniques were described, including both procedures utilizing native semitendinosus tendon with distal attachment left intact as well as with auto- or allo-grafts. However, in part of these techniques, AMRI is not addressed.

Therefore, the aim of this study is to assess the outcomes of the combined quadriceps tendon-bone (QTB) ACLR and MCLR with anteromedial reinforcement performed as described in the published technique: K. Malinowski, K. Hermanowicz, A. Góralczyk, R.F. LaPrade, Medial Collateral Ligament Reconstruction With Anteromedial Reinforcement for Medial and Anteromedial Rotatory Instability of the Knee, Arthrosc. Tech. 8 (2019) e807-e814. https://doi.org/10.1016/j.eats.2019.03.019.

The primary outcome consists of The International Knee Documentation Committee Questionnaire (IKDC) and the Knee injury and Osteoarthritis Outcome Score (KOOS).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic knee medial and anteromedial rotatory instability associated with anterior and rotatory instability after an MCL + ACL injury
* Primary cases

Exclusion Criteria:

* Active inflammation of the knee
* Revision cases
* Additional PLC, PCL or PFJ injuries
* fractures around the knee
* removal of more than ½ of medial or lateral meniscus
* contralateral knee injury
* cartilage damage ICRS grade III or higher
* Non-adherence of the patient to the treatment protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | Before the surgery
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 3 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 6 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 12 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the The International Knee Documentation Committee Questionnaire (IKDC) | At the 24 month of the follow-up.
  Min of 0 max of 87 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | Before the surgery
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 3 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 6 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 12 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome
The functional assessment with the Knee injury and Osteoarthritis Outcome Score | At the 24 month of the follow-up.
  Min of 0 max of 100 points, higher scores mean a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Artromedical Orthopaedic Clinic, Bełchatów, Poland

REFERENCES:
- [Background] Malinowski K, Hermanowicz K, Goralczyk A, LaPrade RF. Medial Collateral Ligament Reconstruction With Anteromedial Reinforcement for Medial and Anteromedial Rotatory Instability of the Knee. Arthrosc Tech. 2019 Jul 18;8(8):e807-e814. doi: 10.1016/j.eats.2019.03.019. eCollection 2019 Aug. PMID 31700776
- [Background] Alm L, Drenck TC, Frings J, Krause M, Korthaus A, Krukenberg A, Frosch KH, Akoto R. Lower Failure Rates and Improved Patient Outcome Due to Reconstruction of the MCL and Revision ACL Reconstruction in Chronic Medial Knee Instability. Orthop J Sports Med. 2021 Mar 15;9(3):2325967121989312. doi: 10.1177/2325967121989312. eCollection 2021 Mar. PMID 33796589
- [Background] Lee DW, Kim JG. Anatomic medial complex reconstruction in serious medial knee instability results in excellent mid-term outcomes. Knee Surg Sports Traumatol Arthrosc. 2020 Mar;28(3):725-732. doi: 10.1007/s00167-019-05367-9. Epub 2019 Apr 17. PMID 30997548
- [Background] Xu H, Kang K, Zhang J, Xin D, Liu W, Jin G, Dong J, Gao S. An anatomical-like triangular-vector ligament reconstruction for the medial collateral ligament and the posterior oblique ligament injury with single femoral tunnel: a retrospective study. J Orthop Surg Res. 2017 Jun 26;12(1):96. doi: 10.1186/s13018-017-0602-3. PMID 28651635
- [Background] Kitamura N, Ogawa M, Kondo E, Kitayama S, Tohyama H, Yasuda K. A novel medial collateral ligament reconstruction procedure using semitendinosus tendon autograft in patients with multiligamentous knee injuries: clinical outcomes. Am J Sports Med. 2013 Jun;41(6):1274-81. doi: 10.1177/0363546513485716. Epub 2013 Apr 26. PMID 23625060
- [Background] Laprade RF, Wijdicks CA. Surgical technique: development of an anatomic medial knee reconstruction. Clin Orthop Relat Res. 2012 Mar;470(3):806-14. doi: 10.1007/s11999-011-2061-1. PMID 21909850
- [Background] Lind M, Jakobsen BW, Lund B, Hansen MS, Abdallah O, Christiansen SE. Anatomical reconstruction of the medial collateral ligament and posteromedial corner of the knee in patients with chronic medial collateral ligament instability. Am J Sports Med. 2009 Jun;37(6):1116-22. doi: 10.1177/0363546509332498. Epub 2009 Mar 31. PMID 19336612
- [Background] Kim SJ, Lee DH, Kim TE, Choi NH. Concomitant reconstruction of the medial collateral and posterior oblique ligaments for medial instability of the knee. J Bone Joint Surg Br. 2008 Oct;90(10):1323-7. doi: 10.1302/0301-620X.90B10.20781. PMID 18827242